CLINICAL TRIAL: NCT02053220
Title: A Phase 1 Clinical Study of Intra-tumoural Injection or Intravenous Infusion of a Group B Oncolytic Adenovirus (ColoAd1) in Patients With Cancer Who Are Candidates for Resection of Primary Tumour
Brief Title: Mechanism of Action Trial of ColoAd1
Acronym: MOA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ColoAd1-1002
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Resectable Colon Cancer; Resectable Non-small Cell Lung Cancer; Resectable Bladder Cancer; Resectable Renal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-tumoural cohort (Experimental)
  Interventions: Biological: Colo-Ad1
- Intra-venous cohort (Experimental)
  Interventions: Biological: Colo-Ad1

INTERVENTIONS:
Biological: Colo-Ad1 — Oncolytic virus

SUMMARY:
To assess the pattern of ColoAd1 viral delivery and viral expression within colon tumour tissue when administered by intra-tumoural injection or within colon, non-small cell lung, bladder and renal cell tumour tissues following ColoAd1 administration by intravenous infusion.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all the following criteria to be eligible for participation:

* Able and willing to provide written informed consent and to comply with the study protocol
* Age ≥ 18 years
* Patients with histologically confirmed resectable colon cancer, NSCLC (squamous and non-squamous), bladder cancer (urothelial cell carcinoma) or RCC (renal cell carcinoma), scheduled for resection of primary tumour and with planned resection of draining lymph nodes for colon cancer
* Diagnostic colonoscopy performed at the study centre (Cohorts A and B only) or a referral centre (Cohort B only) and a report from this colonoscopy available for the study
* Tumour size of 3 cm or more in diameter as estimated during diagnostic colonoscopy for cohorts A and B or by CT-scan for cohorts C, D and E.
* At least 2 weeks since the last dose of any intravenous systemic chemotherapy at time of first administration of ColoAd1
* Recovered to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies.
* Able to undergo surgery with general anaesthesia
* Surgery planned and administration of ColoAd1 feasible within

  * 15 days of planned surgery (following IT administration or following first dose of IV administration) for cohorts A and B
  * 10 - 25 days of first ColoAd1 administration for cohorts C, D and E
* ECOG Performance Status Score of 0 or 1
* Adequate renal function

  * Creatinine ≤ 1.5 mg/dL or calculated creatinine clearance using the Cockcroft-Gault formula ≥ 60 mL/min, or measured creatinine clearance ≥60 mL/min,
  * Absence of clinically significant haematuria on urinalysis: dipstick < 2+
  * Absence of clinically significant proteinuria on urinalysis: dipstick < 2+.
* Adequate hepatic function

  * serum bilirubin <1.5 x ULN
  * AST and ALT ≤ 3 x ULN
* Adequate bone marrow function:

  * ANC ≥ 1.5 x 109/L,
  * platelets ≥ 100 x 109/L,
  * haemoglobin ≥ 90 g/L
* Adequate coagulation tests: INR ≤ 1.5 x ULN;
* For females of childbearing potential (defined as <2 years after last menstruation or not surgically sterile), a negative pregnancy test must be documented prior to enrolment;
* For women who are not postmenopausal (24 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year (e.g., hormonal implants, combined oral contraceptives, vasectomized partner), during the treatment period and for at least 3 months after the last dose of study drug;
* For men: agreement to use a barrier method of contraception during the treatment period and for at least 6 months after the last dose of study drug

Exclusion Criteria for all patients:

Patients who meet any of the following criteria are not eligible for enrolment:

* Rectal tumours; (cohorts A and B);
* An obstructive tumour of the intestine (cohorts A and B only) or of the urinary tract (cohort D);
* Any condition necessitating surgery in less than 8 days (cohorts A or B) or 10 days (cohorts C, D or E);
* Pregnant or lactating (nursing) women;
* Known and/or a history or evidence of significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids at doses higher than dexamethasone 10 mg or equivalent, or other immunosuppressive medications including cyclosporine, azathioprine, interferons, within the past 4 weeks);
* Splenectomy
* Prior allogeneic or autologous bone marrow or organ transplantation
* Active infections requiring antibiotics, physician monitoring, or recurrent fevers >38.0 degrees centigrade associated with a clinical diagnosis of active infection
* Active viral disease, positive serology for HIV, hepatitis B or hepatitis C
* Use of the following anti-viral agents:

  * ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to day 1;
  * or PEG-IFN (within 14 days prior to day 1);
* Administration of an investigational drug within 28 days prior to first dose of ColoAd1
* Major surgery within 4 weeks or radiotherapy within 3 weeks prior to first dose of ColoAd1
* Another primary malignancy within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ)
* Known CNS metastasis
* Inflammatory diseases of the bowel (cohorts A and B only) or any inflammatory disease that may require treatment with corticosteroids.
* Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the drug
* Known allergy to treatment medication or its excipients
* Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Composite measure of viral delivery and spread | Up to Day 25
  To assess the pattern of viral delivery and viral spread of ColoAd1 within tumour tissue when administered either by intra-tumoural injection or by intravenous infusion. Viral delivery and spread will be measured by immunohistochemical staining for ColoAd1 in tumour sections taken from patients. Presence of virus will also be detected by qPCR analysis of tumour tissue.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Madrid Sanchinarro CIOCC, Madrid
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Derived] Garcia-Carbonero R, Salazar R, Duran I, Osman-Garcia I, Paz-Ares L, Bozada JM, Boni V, Blanc C, Seymour L, Beadle J, Alvis S, Champion B, Calvo E, Fisher K. Phase 1 study of intravenous administration of the chimeric adenovirus enadenotucirev in patients undergoing primary tumor resection. J Immunother Cancer. 2017 Sep 19;5(1):71. doi: 10.1186/s40425-017-0277-7. PMID 28923104
- See also: Journal link for MOA study publication — https://jitc.biomedcentral.com/articles/10.1186/s40425-017-0277-7